CLINICAL TRIAL: NCT00306449
Title: Prevention of Weight Gain in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-48
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Weight Gain; Obesity; Overweight
Keywords: Weight gain; obesity; overweight; young adults; lipid disorders; insulin resistance; randomized controled study
MeSH Terms: conditions — Weight Gain; Obesity; Overweight; Lipid Metabolism Disorders; Insulin Resistance

INTERVENTIONS:
Behavioral: Small group seminar-based educational intervention

SUMMARY:
The purpose of the present study is to determine whether weight gain may be prevented by a small group seminar-based two-year educational intervention on healthy lifestyle in freshmen at the Faculté de médecine de l'Université de Sherbrooke.

DETAILED DESCRIPTION:
This is a 2-year randomized, controlled intervention study to test the effectiveness of a small group seminar-based educational intervention on healthy lifestyle to prevent weight gain in young healthy university students.

Hypothesis : We hypothesize that a small group seminar-based educational intervention on healthy lifestyle may prevent weight gain in young healthy adults.

PROTOCOL:

Recrutment of participants : First and second year students will be recruted at the 'Faculté de médecine et des sciences de la santé' of the University of Sherbrooke.

A pre-randomisation visit will be performed to verify eligibility and exclusion criteria and to perform the following:

* Anthropometric measurements (please, see below);
* medical questionnaire;
* physical exam;
* standard questionnaire on dietary and physical activity habits;
* Canadian fitness test (to estimate VO2 max)(www.ecoledudos.uqat.uquebec.ca/chroniquep/03preparationphysique/evaluer/#physitest);
* A fasting blood sample to mesure plasma glucose, insulin, plasma lipids. Serum samples will be stored at -80C for future analyses (adipokines, inflammation markers).

Randomisation: Block randomization according to gender and tertile of BMI of each participant to either the control (no intervention) or intervention (small group seminars) group will be performed once the entire cohort will be recruited at the beginning of the academic year using computer-generated numbers. One investigator will enroll all the study participants and another that will have no contact with the participants will generate the allocation sequence.

Measurements :

A standard questionnaire will be administered to collect the following data: gender, age, study program, medical history, and physical exam results.

Anthropometric measures will be performed at baseline and 3, 6, 12, 18 and 24 months and include:

* Weight (kg),
* height (m) (by standing stadiometre- mean of three measures),
* Waist circumference (cm) (midway between iliac crest and last rib end of a normal expiration - mean of 3 measures),
* lean mass by electrical bio-impedance.

Recording of physical activity : Using a standard questionnaire (Sallis JF et al. Am J Epidemiol 1985;121:91-106) (reported in METs) and performed at 0, 12 and 24 months.

Recording of dietary habits : Standard 3-day food record at 0, 12 and 24 months.

Physical fitness (VO2 max): Canadian Home Fitness Test at 0, 12 and 24 months.

Blood samples (60 ml) at 0 and 24 months: Plasma (15 ml) and serum (15 ml) will be collected after a 8 to 12 hour fast to measure blood glucose; total cholesterol, HDL-cholesterol, total triglycerides (with calculation of LDL-c using the Friedwal formula). Samples will be stored at -80C for future determination of plasma insulin, adipokines and serum inflammatory markers. These analyses will allow us to explore the relationship between weight gain and change in these biological parameters in our study population and to determine whether prevention of weight gain may also be associated with early prevention of metabolic abnormalities associated with obesity.

Intervention:

Small group seminars (10 to 12 students) in the treatment group vs. no specific intervention (other than measurements described above) in the control group. The duration of seminars will be approximatively 30 to 60 minutes and will be given every two weeks for the first two months of follow up and every four weeks for the remaining follow up period, except for summer break (July and August) when seminars will not be given. A multidisciplinary team including endocrinologists, a physical education specialist and a dietician designed the seminars that will be delivered by an endocrinology resident and a physical education graduate student. The first three seminars will be aimed at increasing knowledge on weight gain and its complications, national dietary recommendations (Canadian Food Guide) and exercise categories, expected benefits and recommendations for the maintenance of health. The remaining seminars will be designed to introduce behavioral modification methods using discussion on problem-solving, goal-setting and monitoring strategies. Some seminars will focus on behavioral strategies to maintain a healthy lifestyle during specific periods such as final exams, holidays, winter and vacations. The monitors themselves as well as older students successful at keeping an active lifestyle will be offered as role models to promote a positive image of a healthy lifestyle. Compliance with the intervention will be defined as attending at least 60% of the seminars.

ELIGIBILITY:
Inclusion Criteria:

* Being first or second year in one of the Baccalaureate programs of the Faculté de médecine de l'Université de Sherbrooke.
* Aged between 18 and 30 years old
* BMI between 18 and 30 kg/m2
* Having left parental house less than one year ago

Exclusion Criteria:

* Planned pregnancy or pregnancy occurring during the two-year follow up
* Chronic medical condition that may affect weight present before or occurring during the two-year follow up.
* Use of any medication other than birth control pills.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110
Dates: Start 2002-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Change in weight from baseline between the two groups over a two-year intervention period (0, 3, 6, 12, 18 and 24 months).
Change in BMI from baseline between the two groups over a two-year intervention period (0, 3, 6, 12, 18 and 24 months).

SECONDARY OUTCOMES:
Change in fat free mass (by bioimpedance) over follow up between the two groups.
Change in waist circumference over follow up between the two groups.
Change in non-fat free mass over follow up between the two groups.
Change in dietary intake (by 3-day food records) over follow up between the two groups.
Change in physical activity level (by questionnaire) over follow up between the two groups.
Change in physical fitness level (by the Canadian Home Fitness Test) over follow up between the two groups.
Change in plasma lipid profile (plasma total cholesterol, triglycerides, LDL and HDL cholesterol) over follow up between the two groups.
Change in circulating hormones and inflammatory markers (insulin, leptin, adiponectin, C-reactive protein, Interleukin-6) over follow up between the two groups.
Relation between change in weight and energy intake and expense in the overall cohort.
Relation between change in weight and fitness level in the overall cohort.
Relation between change in weight and metabolic parameters (lipids, hormones and inflammatory markers) in the overall cohort

CONTACTS AND LOCATIONS:
Overall Officials: André C. Carpentier, MD FRCPC, Principal Investigator — Centre de recherche clinique du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre de recherche clinique du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Hivert MF, Langlois MF, Berard P, Cuerrier JP, Carpentier AC. Prevention of weight gain in young adults through a seminar-based intervention program. Int J Obes (Lond). 2007 Aug;31(8):1262-9. doi: 10.1038/sj.ijo.0803572. Epub 2007 Mar 13. PMID 17356531